CLINICAL TRIAL: NCT06575946
Title: Investigation of the Relationship Between the Degree of Hypofunction and Vestibular Tests in Patients With Vestibular Hypofunction
Brief Title: Relationship Between Degree of Hypofunction and Vestibular Tests in Patients With Vestibular Hypofunction
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul Medipol University Hospital (Other)
Responsible Party: Principal Investigator, Ebru Sever, Specialist Physiotherapist, Istanbul Medipol University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: VNG-VESTIBULAR TESTS
Record Dates: First submitted 2024-08-16; First posted 2024-08-28 (Actual); Last update posted 2024-08-28 (Actual); Status verified 2024-08

CONDITIONS: Videonystagmography; Vestibular Assessment
Keywords: Vestibular Hypofunction; Degree of Vestibular Hypofunction; Vestibular Tests

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Vestibular Hypofunction Group (Other)
  Interventions: Diagnostic Test: Vestibular Hypofunction Group

INTERVENTIONS:
Diagnostic Test: Vestibular Hypofunction Group — Demographic information form, vestibular tests, balance tests will be used in the evaluation. The demographic information form includes demographic information (name, surname, gender, smoking, alcohol use, etc.) and clinical conditions (past illnesses and/or surgeries, medications used, whether there is a history of falls, if any, frequency, whether they are afraid of heights and uncomfortable in the dark, etc.). The patients will be diagnosed with videonystagmography (VNG) after the decision of the ENT physician, and their hypofunction levels will be recorded. Vestibular and balance tests will be applied to the patients in the clinical setting. At the end of the study, it will be examined whether there is a relationship between the degree of vestibular hypofunction and the vestibular tests applied in the clinic.

SUMMARY:
Patients with complaints of dizziness and balance problems will be included in the study. Inclusion criteria for the study are; being between the ages of 12-85, having a diagnosis of peripheral vestibular hypofunction. Exclusion criteria from the study are; not being able to communicate, having a diagnosis of central vestibulopathy and having mental disorders. Demographic information form, vestibular tests, balance tests will be used in the evaluation. The demographic information form includes demographic information (name, surname, gender, smoking, alcohol use, etc.) and clinical conditions (past illnesses and/or surgeries, medications used, whether there is a history of falls, if any, frequency, whether they are afraid of heights and uncomfortable in the dark, etc.). The patients will be diagnosed with videonystagmography (VNG) after the decision of the ENT physician, and the degree of hypofunction will be recorded. Vestibular and balance tests will be applied to the patients in a clinical setting. At the end of the study, it will be examined whether there is a relationship between the degree of vestibular hypofunction and the vestibular tests applied in the clinic.

ELIGIBILITY:
Inclusion Criteria:

* Being between 12-85 years old
* Having peripheral vestibular hypofunction
* Having good communication skills and participating in the work willingly

Exclusion Criteria:

* Having wavy vertigo
* Having mental retardation
* Failure to communicate
* Severely limited mobility
* Having acute Meniere's disease
* Having a neurological problem

Ages: 12 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 2000 (Estimated)
Dates: Start 2021-12-01 (Actual); Primary Completion 2022-04-01 (Actual); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Demographic information and data collection form | through study completion, average 2 months
  This form will ask questions about the patient's age, gender, occupation, whether or not they smoke or drink alcohol, accompanying illnesses, previous surgeries, medications they use, daily activity level, history of the disease, onset and type of the disease, whether or not they have fallen in the last year and if so, how many falls, fear of heights, fear of darkness and discomfort with crowds.
Unterberger Test | through study completion, average 2 months
  It is a test that shows which labyrinth is affected and cannot function in peripheral vestibular diseases. The patient makes a counting movement in place 50 times with his eyes closed. If there is a deviation of 45 degrees or more to the right or left after the counting movement, this gives us information that the labyrinth on that side cannot function.
Dynamic Visual Acuity | through study completion, average 2 months
  It is the situation where the visual event is realized clearly while moving. The test is started by passively moving the patient's head in the horizontal plane with a 20° amplitude and 2 Hz speed and the patient starts reading the letters on the Snellen card. The line that can be seen clearly is recorded. The dynamic visual acuity score is the difference between the number of lines on the visual graph when the head is moving passively against the stationary head. In healthy individuals, visual acuity may change by one line in young individuals and by two lines in older individuals. In uncompensated patients, the degree of visual acuity may change by three or two lines in unilateral vestibular losses.
Head Thrust Test | through study completion, average 2 months
  It is a test used to evaluate the function of the vestibulo-ocular reflex (VOR). The head thrust test can be applied in all planes of the semicircular canals. The patient sits on a chair. The physiotherapist or the practitioner stands in front of the patient. The patient is asked to focus on his nose and the patient's head is held and the head is rotated in a horizontal plane with low amplitude and high acceleration. The patient's ability to keep his eyes fixed on the practitioner's nose indicates that there is no problem in the VOR, while corrective saccadic movement indicates that the test is positive.
Timed Balance Tests | through study completion, average 2 months
  Tandem, semitandem, romberg, tek ayak üzerinde durma testleri uygulanacaktır. Bu testler gözler açık ve kapalı olacak şekilde uygulanacaktır. Tek ayak üzerinde durma testleri yumuşak zemin ve sert zeminde olmak üzere iki farklı zeminde yapılacaktır. Testler (sn) olarak ölçülecektir.
Dizziness Handicap Inventory (DHI) | through study completion, average 2 months
  It is used to determine the physical, sensory and functional effects of vestibular system pathologies. Questions 1, 4, 8, 11, 13, 17 and 25 measure physical disability; questions 2, 9, 10, 15, 18, 20, 21, 22 and 23 measure emotional disability; questions 3, 5, 6, 7, 12, 14, 16, 19 and 24 measure functional disability. Each question consists of yes (4 points), no (0 points) and sometimes (2) answers. In scoring the subunits of the inventory, 28 points were accepted as the limit to determine physical disability and 36 points as the limit to determine functional and sensory disability. High scores indicate that the patient's dizziness complaint is at an advanced level.
Tampa Kinesiophobia Scale (TKS) | through study completion, average 2 months
  A 4-point Likert scale (1 = I completely disagree, 4 = I completely agree) is used. It consists of 17 questions. The total score is calculated after reversing items 4, 8, 12 and 16. It gets a total score between 17-68. A high score indicates that kinesiophobia is also high.
Static Posture Assessment with ICS | through study completion, average 2 months
  The Limit of Stability (LOS) program in the balance device called "Otometrics ICS Balance Platform" evaluates the points that the body reaches to maintain balance, the speed of movement and direct control in 8 directions. These directions are; front, right-front, right, right-back, back, left-back, left, left-front. The LOS test measures the maximum distance that an individual can consciously change their center of gravity and extend their body in a certain direction without losing their balance and without taking a step.
Videonystagmography (VNG) | through study completion, average 2 months
  It allows the evaluation of eye movements via cameras sensitive to infrared rays. It is a complex test that allows the examination of the inner ear, including many tests. The test includes; saccade, gaze, tracking, optokinetic, positional tests, Dix Hallpike maneuver and bithermal caloric test. Caloric test is known as the gold standard for the diagnosis of vestibular hypofunction. It reveals the degree, location of hypofunction, whether it is central or peripheral. During the caloric test, thermal stimuli are given and the vestibulo-ocular reflex is evaluated and the pathology is found on which side. 8 liters of air with 50 degrees and 24 degrees temperature, respectively, is sent to the eardrum in 60 seconds with 5-minute rest intervals in both ears. Involuntary eye movements are recorded, calculated and graphed for 120-140 seconds. While evaluating the test result; the onset time of nystagmus, its speed and the possibility of suppression with fixation are examined.

CONTACTS AND LOCATIONS:
Overall Officials: Ebru SEVER, Master's, Principal Investigator — Physiotherapy and Rehabilitation; Gamze KILIÇ, Asst. Prof., Study Director — Physiotherapy and Rehabilitation; Gönül ERTUNÇ GÜLÇELİK, Asst. Prof., Study Director — Physiotherapy and Rehabilitation
Locations (1):
- Güneşli Erdem Hospital, Bağcılar, Güneşli, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No